CLINICAL TRIAL: NCT03576274
Title: Effectiveness of the Combined Technology-enhanced Home Exercise Program and Other Non-pharmacological Interventions on Fatigue, Physical Function and Well-being Among Cancer Survivors
Brief Title: Combined Technology Enhanced Home Exercise Program and Other Non-pharmacological Intervention for Cancer Survivors
Acronym: TEHEplus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Johns Hopkins University (Other); Oncology Nursing Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: J1876; IRB00154198 (Other: JHM IRB)
Record Dates: First submitted 2018-06-07; First posted 2018-07-03 (Actual); Results first posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Cancer-related Problem/Condition; Exercise; Acupressure
Keywords: Cancer related fatigue; Exercise; biomarkers; Auricular Point Acupressure
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Technology Enhanced Home Exercise only (Experimental): Participants in TEHE group will receive a combined technology and home exercise program. Participants will schedule an online meeting with the research team for exercise goal setting and preference. Participants will receive a daily symptoms survey. They will receive, reminder, motivation message and physical performance feedback though the mobile phone application.
  Interventions: Behavioral: Technology Enhanced Home Exercise (TEHE)
- Technology Enhanced Home Exercise plus (Experimental): In additional to the TEHE program, participants will receive auricular point acupressure (APA) training on how to locate the ear points, place the seeds and apply the pressure on the seed.
  Participants will be instructed to press the tape and seeds covering each ear point for 3 minutes per time with a 2-second pause in between pressing, three times daily (morning, afternoon and evening: 9 minutes total).
  The tape and seeds will remain on ear points for 5 days. Participants will be instructed to remove both at the end of the 5th day.
  Interventions: Behavioral: Technology Enhanced Home Exercise (TEHE); Behavioral: Auricular Point Acupressure (APA)
- Technology Enhanced Home Exercise-Mindfulness intervention (Experimental): In addition to the TEHE program, the TEHE+MBI group will receive a audio-recording of a mindfulness-based body scan.
  During the weekly study visit: Participants will be instructed to listen to the recorded mindfulness-based body scan in the morning and before bedtime.
  At home: Participants will be asked to listen to this audiotape daily in the morning and before bedtime.
  Interventions: Behavioral: Technology Enhanced Home Exercise (TEHE); Behavioral: Mindfulness body scan (MBI)
- Control (usual care) (No Intervention): The control group will receive instructions on how to use the physical activity tracker and mEMA application. Participants will be asked to meet with a research team member weekly to discuss their fatigue experience and receive general information about fatigue management.
- Auricular Point Acupressure only (Active Comparator): Participants will receive auricular point acupressure (APA) training on how to locate the ear points, place the seeds and apply the pressure on the seed.
  Participants will be instructed to press the tape and seeds covering each ear point for 3 minutes per time with a 2-second pause in between pressing, three times daily (morning, afternoon and evening: 9 minutes total).
  The tape and seeds will remain on ear points for 5 days. Participants will be instructed to remove both at the end of the 5th day.
  Interventions: Behavioral: Auricular Point Acupressure (APA)

INTERVENTIONS:
Behavioral: Technology Enhanced Home Exercise (TEHE) — A 12 week program including one 60-minute goal setting and exercise training program and follow up phone calls.
  Arms: Technology Enhanced Home Exercise only; Technology Enhanced Home Exercise plus; Technology Enhanced Home Exercise-Mindfulness intervention
Behavioral: Auricular Point Acupressure (APA) — A non invasive complementary method to provide pressure on the ear points.
  Arms: Auricular Point Acupressure only; Technology Enhanced Home Exercise plus
Behavioral: Mindfulness body scan (MBI) — The open, nonjudgmental attention to move one's attention calmly to the different part of the body
  Arms: Technology Enhanced Home Exercise-Mindfulness intervention

SUMMARY:
A 12 weeks technology enhanced home exercise (TEHE) program using mobile technologies that provide immediate feedback and send reminder messages to improve exercise motivation is developed. Investigators combine this TEHE program with techniques including auricular point pressure (APA) and brief mindfulness body scan (MBI). This study will examine the feasibility of the TEHE program and combined programs, and ascertain the effect of TEHE program alone, the combined programs on fatigue and biological markers among cancer survivors.

Main Research Variable(s): The independent variables are the 12-week program of TEHE alone, APA alone, combined APA and TEHE (TEHEplus) and combined MBI and TEHE (TEHE-MBI). Outcome variables are fatigue, physical activity, contributing factors of fatigue and biomarkers.

Design: Repeated measures randomized controlled trial. Setting: Participants will be recruited through the Comprehensive Cancer Center, Johns Hopkins University.

Sample: Participants diagnosed with non-metastatic solid tumor cancer; who had completed all primary cancer treatment (surgery, chemotherapy, and radiation therapy )within at least 3 months OR non-metastatic prostate cancer completed all primary cancer treatment and have hormone therapy for at least 6 month, OR participants diagnosed with solid tumor cancer; who are receiving immunotherapy for at least 3 months before enrollment, aged 21 years or older, experiencing fatigue in the past 7 days on average of ≥ 3/10, able to participate in a moderate-intensity exercise training program, self-report ability to complete the 6 min walk test with a perceived exertion of 3 or below, and can communicate in English.

Methods: Participants who meet the inclusion criteria will be randomly assigned to the TEHE only, APA only or TEHEplus or TEHE-MBI or control group. All exercise groups (TEHE) will be offered a 12-week exercise program through an online communication. In additional to the TEHE, the TEHEplus group will receive an instruction on how to apply the pressure on the ear points through online meeting/communication. The TEHE-MBI group will perform 5 min mindfulness body scan daily. The control (usual care) group will report participant's fatigue level daily. At the end of week 12, participants will answer open-ended questions about participant's opinions on the programs. Fatigue will be assessed and blood will be drawn before and after the program.

DETAILED DESCRIPTION:
Home-based exercise interventions have a significant effect on fatigue; however, motivation and intervention compliance are the main challenges. The use of personalized exercise and immediate feedback though smartphome communication has been found to increase motivation. We developed a 12 weeks technology enhanced home exercise (TEHE) program using mobile technologies that provide immediate feedback and sends reminder messages to improve exercise motivation. Moreover, to enhance the effectiveness of exercise, we combine this TEHE program with techniques--auricular point pressure and brief mindfulness body scan--, which have been found to affect fatigue and physical activities. The Auricular Point Acupressure (APA) and Mindfulness Based Intervention (MBI) may enhance the effect of exercise on fatigue; however, the feasibility and effectiveness of this combination have not been tested. This study will examine the feasibility of the TEHEplus program and ascertain the effect of TEHE program alone, APA alone, the TEHEplus program and the TEHE-MBI program on fatigue among cancer survivors and cancer patients receiving immunotherapy. In addition we will explore peripheral and central markers (e.g., Phosphorous levels) of cancer-related fatigue using magnetic resonance spectroscopy (MRS). This study will also investigate whether specific types of fatigue (e.g., physical fatigue, cognitive fatigue) will have different levels of these peripheral and central energy markers).

Conceptual Framework: The biopsychosocial model will be used. Main Research Variable(s): The independent variables are the 12-week program of TEHE alone, APA alone, combined APA and TEHE (TEHEplus) and combined MBI and TEHE (TEHE-MBI). Outcome variables are fatigue, physical activity, contributing factors of fatigue (depressive symptom, anxiety, sleep, relationship with others), and biomarkers.

Design: Repeated measures randomized controlled trial design. Setting: Participants will be recruited through the Comprehensive Cancer Center, Johns Hopkins University.

Sample: Participants diagnosed with non-metastatic solid tumor cancer; who had completed all primary cancer treatment (surgery, chemotherapy, and radiation therapy )within at least 3 months OR non-metastatic prostate cancer completed all primary cancer treatment and have hormone therapy for at least 6 month, OR participants diagnosed with solid tumor cancer; who are receiving immunotherapy for at least 3 months before enrollment, aged 21 years or older, experiencing fatigue in the past 7 days on average of ≥ 3/10, able to participate in a moderate-intensity exercise training program, self-report ability to complete the 6 min walk test with a perceived exertion of 3 or below, and can communicate in English.

Methods: Participants who meet the inclusion criteria will be randomly assigned to the TEHE only, APA only, TEHEplus or TEHE-MBI or control (usual care) group. All exercise groups will be offered a 12-week exercise program. The program will based on personal exercise preference and physical activity goals to reach moderate intensity based on readings from a heart rate monitor and exertion level. Activity/steps will be monitored daily using the FitBit Charge. Reminders to exercise will be sent to the patient through a mobile phone application based on the participants' personal schedule and frequency. In additional to the TEHE, the APA only, and the TEHEplus group will receive an instruction on how to apply the pressure on the ear points through the online meeting and mobile application. The TEHE-MBI group will perform 5 min of mindfulness body daily. The control (usual care) group will report their fatigue level daily and attend weekly meetings with the researcher to discuss fatigue. At the end of week 12, in addition to the questionnaires, participants will answer open-ended questions about their opinions on the program. Fatigue will be assessed and blood will be drawn before and after the program. Participants who enrolled in the sub-study will be scheduled for a visit for an MRS before the exercise intervention.

2. Objectives (include all primary and secondary objectives)

Purpose/Specific Aims:

The study primary aims are to (1) test the feasibility of a 12-week technology-enhanced home exercise (TEHE) program and combined technology-enhanced home exercise and Auricular Point Acupressure (TEHE plus) program among cancer survivors; (2) to determine the effect of the TEHE plus program on fatigue, physical activity and serum biomarkers (Heat Shock Protein 90 and Brain-Derived Neurotrophic Factor) compared to the control (usual care) group.

The secondary aims are to (3) compare the effect of the TEHE only, TEHE plus, APA only, combined MBI and TEHE on fatigue and physical activity; and (4) determine the change in serum biomarkers at week 12 compared to baseline in the TEHE only, TEHE plus, APA only, MBI+TEHE, and control (usual care) groups (5) explore the associations of muscle and brain energetic markers using magnetic resonance spectroscopy (MRS) with fatigue symptoms of cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with non-metastatic solid tumor cancer; who had completed all primary cancer treatment (surgery, chemotherapy, and radiation therapy )within at least 3 months OR non-metastatic prostate cancer completed all primary cancer treatment and have hormone therapy for at least 6 month, OR participants diagnosed with solid tumor cancer; who are receiving immunotherapy for at least 3 months before enrollment
* aged 21 years or older, experiencing fatigue in the past 7 days on average of ≥ 3/10
* able to participate in a moderate-intensity exercise training program (self-report ability to complete the 6 min walk test with a perceived exertion of 3 or below)
* able to communicate in English.

Exclusion Criteria:

* diagnosed with comorbidities, such as cardiovascular, lung, kidney, liver, or thyroid diseases
* have an active infection (e.g., fever, localized redness, swelling, sinus congestion)
* diagnosed with a psychological disorder (e.g., suicidal or homicidal tendencies, extreme anxiety or depression)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nada Lukkahatai, PhD, Principal Investigator — Johns Hopkins School of Nursing
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Lukkahatai N, Benjasirisan C, Shen A, Li J, Allgood S, Thomas F, Karyukin A, Sheng JY, Engle J, Lee TY, Saligan LN. Combined technology-enhanced home exercise and acupressure (TEHEplus) program on symptoms among cancer patients receiving immunotherapy: a feasibility study. BMC Cancer. 2025 Oct 1;25(1):1481. doi: 10.1186/s12885-025-14887-2. PMID 41034793

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Johns Hopkins-affiliated hospitals (Sibley Memorial, Bayview, and JHH) and via social media, co-investigator referrals, and JHU-ICTR MyChart messages. Flyers and bookmarks directed potential participants to a REDCap screening survey. Recruitment included clinical settings and online platforms. Participants were contacted by the PI or research staff.
Groups:
- Technology Enhanced Home Exercise Plus: In additional to the TEHE program, participants will receive auricular point acupressure (APA) training on how to locate the ear points, place the seeds and apply the pressure on the seed.
  Participants will be instructed to press the tape and seeds covering each ear point for 3 minutes per time with a 2-second pause in between pressing, three times daily (morning, afternoon and evening: 9 minutes total).
  The tape and seeds will remain on ear points for 5 days. Participants will be instructed to remove both at the end of the 5th day.
  Technology Enhanced Home Exercise (TEHE): A 12 week program including one 60-minute goal setting and exercise training program and follow up phone calls.
  Auricular Point Acupressure (APA): A non invasive complementary method to provide pressure on the ear points.
- Technology Enhanced Home Exercise-Mindfulness Intervention: In addition to the TEHE program, the TEHE+MBI group will receive a audio-recording of a mindfulness-based body scan.
  During the weekly study visit: Participants will be instructed to listen to the recorded mindfulness-based body scan in the morning and before bedtime.
  At home: Participants will be asked to listen to this audiotape daily in the morning and before bedtime.
  Technology Enhanced Home Exercise (TEHE): A 12 week program including one 60-minute goal setting and exercise training program and follow up phone calls.
  Mindfulness body scan (MBI): The open, nonjudgmental attention to move one's attention calmly to the different part of the body
- Auricular Point Acupressure Only: Participants will receive auricular point acupressure (APA) training on how to locate the ear points, place the seeds and apply the pressure on the seed.
  Participants will be instructed to press the tape and seeds covering each ear point for 3 minutes per time with a 2-second pause in between pressing, three times daily (morning, afternoon and evening: 9 minutes total).
  The tape and seeds will remain on ear points for 5 days. Participants will be instructed to remove both at the end of the 5th day.
  Auricular Point Acupressure (APA): A non invasive complementary method to provide pressure on the ear points.
Period: Overall Study
Arm/Group | Technology Enhanced Home Exercise Only | Technology Enhanced Home Exercise Plus | Technology Enhanced Home Exercise-Mindfulness Intervention | Control (Usual Care) | Auricular Point Acupressure Only
Started | 22 | 23 | 21 | 22 | 22
Completed | 14 | 18 | 16 | 13 | 13
Not Completed | 8 | 5 | 5 | 9 | 9
Not completed — Lost to Follow-up | 3 | 2 | 3 | 1 | 3
Not completed — Withdrawal by Subject | 5 | 3 | 2 | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Technology Enhanced Home Exercise Only | Technology Enhanced Home Exercise Plus | Technology Enhanced Home Exercise-Mindfulness Intervention | Control (Usual Care) | Auricular Point Acupressure Only | Total
Number analyzed (Participants) | 22 | 23 | 21 | 22 | 22 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (12) | 61 (12) | 61 (12) | 60 (13) | 58 (13) | 60 (12)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 9 | 9 | 10 | 9 | 8 | 45
  Sex: Male | 12 | 14 | 11 | 13 | 14 | 64
  Sex: Not reported | 1 | 0 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 1 | 2 | 8
  Not Hispanic or Latino | 16 | 17 | 16 | 19 | 18 | 86
  Unknown or Not Reported | 4 | 5 | 3 | 2 | 2 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 2 | 1 | 2 | 1 | 6
  White | 18 | 20 | 20 | 18 | 19 | 95
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 1 | 1 | 5
Education [Count of Participants; unit: Participants]
  High school and below | 1 | 1 | 1 | 0 | 0 | 3
  Some college/associate degree | 1 | 4 | 2 | 8 | 5 | 20
  Bachelor's degree or higher | 19 | 18 | 18 | 11 | 15 | 81
  Not reported | 1 | 0 | 0 | 3 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Fatigue on the Patient-reported Outcomes Measure Information System (PROMIS-F) From Baseline to Week 12 (Post-intervention)
Description: Fatigue will be measured by the self-report questionnaire including 1) the PROMIS-F, self self-report measure that assesses fatigue over the past 7 days. Score range 8-40 with higher score indicating worse fatigue.
Time Frame: Baseline and week 12 (post-intervention)
Population: Participants with data collected at both baseline and post-intervention are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Technology Enhanced Home Exercise Only | Technology Enhanced Home Exercise Plus | Technology Enhanced Home Exercise-Mindfulness Intervention | Control (Usual Care) | Auricular Point Acupressure Only
Number analyzed (Participants) | 14 | 18 | 16 | 13 | 13
score on a scale | -3.8 (11.0) | -7.9 (19.8) | -5.8 (13.3) | -3.2 (9.2) | -3.3 (9.3)

2. Secondary Outcome: Change in Right-hand Skeletal Muscle Strength, Measured Using a Hand-held Dynamometer, From Baseline to Week 12 (Post-intervention)
Description: Skeletal muscle strength was assessed by averaging the maximum force exerted across three trials for each hand using a hand-held dynamometer, with results recorded in pounds (lb).
Time Frame: Baseline and week 12 (post-intervention)
Population: Participants with data collected at both baseline and post-intervention are reported.
Measure: Mean (Standard Error); unit: pounds (lb)
Arm/Group | Technology Enhanced Home Exercise Only | Technology Enhanced Home Exercise Plus | Technology Enhanced Home Exercise-Mindfulness Intervention | Control (Usual Care) | Auricular Point Acupressure Only
Number analyzed (Participants) | 3 | 10 | 3 | 3 | 4
pounds (lb) | 9.9 (33.2) | -2.5 (10.2) | 2.8 (2.1) | -3.1 (6.6) | -0.4 (3.6)

3. Secondary Outcome: Change in Left-hand Skeletal Muscle Strength, Measured Using a Hand-held Dynamometer, From Baseline to Week 12 (Post-intervention)
Description: as for outcome 2
Time Frame: Baseline and week 12 (Post-intervention)
Population: Participants with data collected at both baseline and post-intervention are reported.
Measure: Mean (Standard Deviation); unit: pounds (lb)
Arm/Group | Technology Enhanced Home Exercise Only | Technology Enhanced Home Exercise Plus | Technology Enhanced Home Exercise-Mindfulness Intervention | Control (Usual Care) | Auricular Point Acupressure Only
Number analyzed (Participants) | 3 | 10 | 3 | 3 | 4
pounds (lb) | 4.4 (17.6) | -0.7 (12.0) | 3.0 (1.3) | -2.4 (11.6) | 19.8 (45.7)

4. Secondary Outcome: Change in Brain Derived Neurotrophic Factors Between Baseline to Week 12 (Post-intervention)
Description: Peripheral venous blood was collected in serum tubes for plasma BDNF analysis both before and after the intervention. Plasma level of Brain Derived Neurotrophic Factors measured in ug/ml
Time Frame: Between baseline and week 12 (post-intervention)
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Technology Enhanced Home Exercise Only | Technology Enhanced Home Exercise Plus | Technology Enhanced Home Exercise-Mindfulness Intervention | Control (Usual Care) | Auricular Point Acupressure Only
Number analyzed (Participants) | 22 | 23 | 21 | 22 | 22
ug/ml | -4945.7 (8777.9) | -3971.3 (9551.5) | -106.5 (1078.8) | -2013.3 (5807) | -2912.8 (13780)

5. Secondary Outcome: Change in Heat Shock Protein Level Measured in pg/ml From Baseline to Week 12 (Post-intervention)
Description: Plasma level of Heat Shock Protein 90 (HSP90) measured in ug/ml from baseline to Week 12 (post-intervention)
Time Frame: Baseline and week 12 (post-intervention)
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Technology Enhanced Home Exercise Only | Technology Enhanced Home Exercise Plus | Technology Enhanced Home Exercise-Mindfulness Intervention | Control (Usual Care) | Auricular Point Acupressure Only
Number analyzed (Participants) | 22 | 23 | 21 | 22 | 22
ug/ml | -325.6 (860.9) | -106.5 (1078.8) | 3.39 (859.1) | -297.0 (753.1) | -396.7 (1465.3)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Arm/Group | Technology Enhanced Home Exercise Only | Technology Enhanced Home Exercise Plus | Technology Enhanced Home Exercise-Mindfulness Intervention | Control (Usual Care) | Auricular Point Acupressure Only
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23 | 0/21 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/21 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 1/23 | 0/21 | 0/22 | 0/22
OTHER ADVERSE EVENTS (reported when occurring in more than 4.35% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Technology Enhanced Home Exercise Only (N=22) | Technology Enhanced Home Exercise Plus (N=23) | Technology Enhanced Home Exercise-Mindfulness Intervention (N=21) | Control (Usual Care) (N=22) | Auricular Point Acupressure Only (N=22)
Wrist discomfort on the non-dominant wrist (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 0 | 0 — Patient reported wrist discomfort on the non-dominant wrist with no rash, redness, and/or swelling.

LIMITATIONS AND CAVEATS:
The study's limitations include a small sample size and low statistical power, as it was designed as a pilot to assess feasibility rather than detect statistically significant effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT03576274/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT03576274/ICF_001.pdf